CLINICAL TRIAL: NCT00985582
Title: Antiviral Treatment in Adults and Children With Novel Influenza A (H1N1) Respiratory Tract Infection - a Clinical, Virological and Pharmacokinetic Study.
Brief Title: Antiviral Therapy for Influenza A H1N1
Acronym: SEA032
Status: Completed | Type: Observational
Sponsor: South East Asia Infectious Disease Clinical Research Network (Network)
Collaborators: Wellcome Trust (Other)
Responsible Party: Prof. Jeremy Farrar FRCP Dphil / Principal Investigator, Oxford University Clinical Research Unit, Ho Chi Minh City, Vietnam
Other Study IDs: SEA032
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Influenza A Virus Infection
Keywords: Influenza A Virus (H1N1)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swabs, throat swabs, nasopharyngeal aspirates, rectal swabs, urine, blood, will be obtained for virological analyses, according to the age group specific study schedules
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aims of this study are to characterise the clinical efficacy and virological clearance dynamics of orally administered oseltamivir in patients with influenza caused by novel influenza A(H1N1). This research will also contribute to enhancing research capacity in affected countries.

The objectives are to assess the:

* viral replication levels over time in affected patients
* antiviral efficacy of oral oseltamivir
* patterns and compartments of viral shedding, tissue distribution
* innate inflammatory response and relation to viral replication
* kinetics of antibody response
* antiviral sensitivity of influenza viruses at baseline and during oseltamivir treatment using in vitro and molecular methods
* pharmacokinetic characteristics of oseltamivir and oseltamivir carboxylate
* all cause in hospital mortality
* clinical and radiological features, disease course and outcome
* length of stay in hospital
* risk factors associated with development of severe disease and death

DETAILED DESCRIPTION:
Any patient over 1 year of age who presents to a participating institution with confirmed influenza A and who meets the study inclusion/exclusion criteria may be approached for informed consent. Choice of antiviral is up to the study physician. Children aged 1-6 years and asthmatics should receive oseltamivir. The weight- and age-adjusted dosage used will be that approved for treatment of uncomplicated seasonal influenza, and doses will be administered twice daily for 5 days for patients with normal renal function. All patients who are clinical and/or virologic failures at day 5 will be treated for an additional 5 days of antivirals. After coming off antiviral therapy patients can be discharged at day 10 if deemed ready by study physicians and they are virologically negative.

During the course of treatment study evaluations will be performed to determine primary efficacy end points including viral clearance on Day 5 on all collected nasopharyngeal samples, assessed by RT PCR for novel H1N1 influenza AND no clinical features of clinical failure. Evaluations will also be performed to determine secondary viral, serological, clinical efficacy, safety and pharmacokinetic endpoints.

Patients will be followed up for up to 6 months after discharge for a clinical assessment, pulmonary function and outcome of pregnancy.

The protocol will be reviewed after 6 months from starting or after 100 patients with Influenza A are recruited.

ELIGIBILITY:
Inclusion Criteria:

* Adults, including pregnant and breast feeding women, and Children aged ≥ 12 months when first seen with an acute febrile respiratory tract illness (ARI) of any severity and influenza A, virologically proven on a respiratory specimen according to hospital procedure, which is suspected to be novel influenza A(H1N1)
* A positive influenza A H1 swine screening reverse transcriptase polymerase chain reaction (RT PCR) or conventional PCR assay on one respiratory specimen : NPA, NP swab, nasal wash, nasal swab and throat swab
* Underlying illnesses including HIV
* Prescribed oseltamivir prior to presentation

Exclusion Criteria:

* Lack of informed consent

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a single arm clinical and virological study assessing the use of oral oseltamivir or other agents in the treatment of patients with novel influenza A(H1N1) infection.
  Any patient over 1 year of age with confirmed novel influenza A(H1N1) in whom appropriate informed consent to collect data and samples is obtained. The protocol will be reviewed after 6 months from starting or after 100 patients with new influenza A(H1N1) are recruited.
Sampling Method: Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Viral clearance on Day 5 on all collected nasopharyngeal samples, assessed by RT PCR for new influenza A(H1N1) | 12 months

SECONDARY OUTCOMES:
Viral clearance on Day 1, 2, 3, 4, 5 (H1N1) on nose and throat swab, assessed by RT PCR. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Farrar, MD, Principal Investigator — Oxford University Clinical Research Unit Ho Chi Minh City Vietnam
Locations (1):
- National Institute for Infectious and Tropical Diseases (NIITD), Viet Nam, Hanoi, Vietnam

REFERENCES:
- [Background] Lackenby A, Thompson CI, Democratis J. The potential impact of neuraminidase inhibitor resistant influenza. Curr Opin Infect Dis. 2008 Dec;21(6):626-38. doi: 10.1097/QCO.0b013e3283199797. PMID 18978531
- [Background] Ferraris O, Lina B. Mutations of neuraminidase implicated in neuraminidase inhibitors resistance. J Clin Virol. 2008 Jan;41(1):13-9. doi: 10.1016/j.jcv.2007.10.020. Epub 2007 Dec 11. PMID 18055254
- [Background] Shiraishi K, Mitamura K, Sakai-Tagawa Y, Goto H, Sugaya N, Kawaoka Y. High frequency of resistant viruses harboring different mutations in amantadine-treated children with influenza. J Infect Dis. 2003 Jul 1;188(1):57-61. doi: 10.1086/375799. Epub 2003 Jun 23. PMID 12825171
- [Background] Hurt AC, Ho HT, Barr I. Resistance to anti-influenza drugs: adamantanes and neuraminidase inhibitors. Expert Rev Anti Infect Ther. 2006 Oct;4(5):795-805. doi: 10.1586/14787210.4.5.795. PMID 17140356
- [Background] Dutkowski R, Thakrar B, Froehlich E, Suter P, Oo C, Ward P. Safety and pharmacology of oseltamivir in clinical use. Drug Saf. 2003;26(11):787-801. doi: 10.2165/00002018-200326110-00004. PMID 12908848